CLINICAL TRIAL: NCT05004922
Title: The Correlation Between the Site of Embryo Transfer and the Site of Gestational Sac and Placental Implantation
Brief Title: Site of Embryo Transfer in Intracytoplasmic Sperm Injection
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: National Research Centre, Egypt (Other)
Responsible Party: Principal Investigator, Sherif Elsirgany, Researcher ,Family Planning and Reproductive Health Department, National Research Centre, Egypt
Other Study IDs: ICSI
Record Dates: First submitted 2019-02-03; First posted 2021-08-13 (Actual); Last update posted 2021-08-13 (Actual); Status verified 2021-08

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ICSI in upper cavity: Embryo transfer into the upper cavity
  Interventions: Other: Embryo transfer into upper cavity
- ICSI in midcavity: Embryo transfer into the midcavity
  Interventions: Other: Embryo transfer into midcavity

INTERVENTIONS:
Other: Embryo transfer into upper cavity — Transfer of embryos in upper cavity
  Other Names: Gestational sac site after embryo transfer
  Groups: ICSI in upper cavity
Other: Embryo transfer into midcavity — Transfer of embryos in mid cavity
  Other Names: Gestational sac site after embryo transfer
  Groups: ICSI in midcavity

SUMMARY:
The technique of embryo transfer is thought to affect the implantation and pregnancy rate .At present, the implantation site can be estimated from the location of the very early gestational sac by transvaginal ultrasound.

DETAILED DESCRIPTION:
Many authors claimed that an increase in implantation and pregnancy rates has been reported to occur when embryos are transferred to the central area of the uterine cavity but there are no studies about the implantation site after using this type of transfer.

ELIGIBILITY:
Inclusion Criteria:

* 1- AVF uterus. 2- BMI less than 30

Exclusion Criteria:

* 1- RVF uterus. 2- BMI more than 30.

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — women with infertility who will undergo ICSI
Study Population: infertile women
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2021-09-01 (Estimated); Primary Completion 2022-01-01 (Estimated); Study Completion 2022-02-01 (Estimated)

PRIMARY OUTCOMES:
number of women who will get pregnant in each group | within one month
  how many women will get pregnant after ICSI in every group

CONTACTS AND LOCATIONS:
Overall Officials: Sherif Elsirgany, M.D, Principal Investigator — Researcher, Family planning and Reproductive Health Department, NRC, Egypt

IPD SHARING:
Plan to Share IPD: Undecided